CLINICAL TRIAL: NCT06469723
Title: Protocol for Inpatient Nursing Frailty Assessment (INFA): Comprehensive Geriatric Assessment and Multidisciplinary Intervention for Frail Hospitalised Older Adults
Brief Title: Protocol for Inpatient Nursing Frailty Assessment (INFA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Geriatric Education and Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/00937
Record Dates: First submitted 2024-05-06; First posted 2024-06-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-07

CONDITIONS: Functional Status; Frailty
Keywords: INFA; Inpatient Nursing Frailty Assessment; Consolidated Framework for Implementation Research; CFIR; Functional Status; Healthcare utilization; Cost Effectiveness Analysis
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Two General Medicine (GM) wards and two General Surgery (GS) wards will be used for the study.
  One GM and one GS ward will be designated as INFA intervention wards while the remaining two wards will be designated as control.
  Participants will be randomly sorted into either of the wards and outcome data will be collected from the participants at three timepoints: Baseline (Admission), discharge, and 6-months post discharge.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INFA Intervention (Experimental): Participants sorted into this arm will receive care under the INFA program, which includes standard care, along with early detection of geriatric syndromes or symptoms using the INFA screening tool. This will include potential early referrals to allied health professionals, care plans, and comprehensive early discharge planning and systematic follow-ups.
  Interventions: Other: INFA Program
- Standard Care - Control (No Intervention): Participants sorted into this arm will continue to receive standard care in the wards.

INTERVENTIONS:
Other: INFA Program — Participants will be screened using the INFA Screening tool, comprising of assessments for multiple domains that are part of existing routine admission nursing assessments, including functional decline, delirium, recurrent falls, self-reported hearing and visual impairment questionnaires, malnutrition risk, oral health, and dysphagia screening. Nurse-led protocols will be done to address each identified geriatric syndrome.
  Participants with complex cases (defined as delirium and/or high-risk falls) will be referred to the GeriCARE service, with capabilities for performing comprehensive geriatric assessment (CGA) guiding discharge planning. Referrals to geriatricians can be initiated whenever necessary, facilitating access to specialised geriatric medical expertise.
  Participants will also receive comprehensive discharge planning and systematic follow-up procedures, done by ward resource nurses.
  Arms: INFA Intervention

SUMMARY:
Background:

Frailty confers greater risks of negative health outcomes in hospitalised older adults. To improve care for this vulnerable population, Comprehensive Geriatric Assessment (CGA) is recommended for frail older persons. However, implementing CGA outside of specialised geriatrician-led settings is limited, and few care models use frailty to identify and target older persons for CGA in the hospital-wide context.

The Inpatient Nursing Frailty Assessment (INFA) programme is a CGA-based care model that targets frail older adults acutely admitted to the hospital under non-geriatrician care. The INFA collects information from routine admission assessments by ward nurses, identifying CGA domains of functional decline, delirium, falls, sensory impairment, nutrition, oral health, and swallowing. The CGA allows earlier identification of health issues and development of a personalised care plan, which directs patients to resources that mitigate the risks of functional decline. Resources include nurse-initiated interventions, multidisciplinary team care, discharge planning, community care referrals, and specialist geriatric medicine reviews.

Methods:

The investigators aim to evaluate the INFA programme over two phases: pre-implementation and implementation. The updated CFIR including its Outcomes Addendum is the framework guiding both phases in the evaluation of effectiveness and implementation. The investigator's hybrid type 2 effectiveness-implementation study design is anchored in this framework. During pre-implementation, the investigators will evaluate the determinants of implementation success and subsequently refine implementation strategies. In the implementation phase, the investigators apply a quasi-experimental approach with intervention and control groups to examine the effects of the INFA intervention compared to usual care. Study participants are patients admitted to medical and surgical wards and are not receiving geriatric care. Individuals are aged 65 years and above and mild to moderately frail (CFS score 4-6). Implementation research in this phase aims to evaluate implementation outcomes. The primary outcome is activities of daily living at six months post-discharge. Secondary outcomes include length of stay, healthcare utilisation including readmissions and ED visits, quality-of-life, and cost-effectiveness.

Discussion:

The study's overall goal is to enhance the quality of care for frail older adults during their hospital stay, leading to improved functional outcomes.

DETAILED DESCRIPTION:
The Inpatient Nursing Frailty Assessment (INFA) programme is a Comprehensive Geriatric Assessment (CGA)-based care model that targets frail older adults acutely admitted to the hospital under non-geriatrician care.

Briefly, the INFA programme includes: (1) A comprehensive geriatric syndrome screening tool, merging multiple assessment areas into a streamlined Epic template. This unified system optimises patient data capture and monitoring, promoting early detection of geriatric syndromes; (2) Nurse-led intervention protocols, offering detailed strategies for managing identified geriatric syndromes. This development equips nurses with skills to address complex needs of frail adults, through additional training and supervision; (3) An improved referral process for complex cases to specialist Geriatric nursing and medical care; and (4) Comprehensive early discharge planning and systematic follow-up procedures involving both internal hospital personnel and external community service teams.

This study aims to use the updated Consolidated Framework for Implementation Research (CFIR) including its Outcomes Addendum to guide the evaluation of the effectiveness and implementation of the INFA programme over two phases: pre-implementation and implementation.

In the pre-implementation phase, a detailed written description of the INFA care model will be produced. We will also create a logic model to describe the activities, outputs and outcomes of INFA will be constructed and a theory of change model to explain the causal pathways linking them will be developed. The investigators will engage implementors (healthcare professionals) through focus group discussions (FGDs) and in-depth interviews (IDIs) to understand their perspectives on various contextual factors to implementing the INFA program, thereby enhancing the chances of successful and sustained implementation.

Each participant will attend either a FGD or IDI covering the barriers and facilitators, framed as CFIR determinants, that influence the acceptability, feasibility, and adoptability of the INFA programme, prior to implementation.

The investigators will identify strategies from the Expert Recommendations for Implementing Change compilation (ERIC) before using the CFIR-ERIC matching tool to select implementation strategies to address CFIR-identified contextual barriers based on the implementer's views.

In the implementation phase, the investigators will apply a quasi-experimental pretest-posttest design with intervention and control groups to examine the effects of the INFA intervention compared to standard care.In the implementation phase, the investigators will apply a quasi-experimental pretest-posttest design with intervention and control groups to examine the effects of the INFA intervention compared to standard care. There will be one control and one intervention ward in General Medicine and General Surgery wards. Evaluations on the primary outcome of interest - Functional status - will occur at baseline (admission), discharge, and six months post-discharge. Secondary outcomes and cost-effectiveness analysis will also be collected and analyzed during this study.

Importantly, the implementation phase involves implementation research. The investigators will evaluate the degree of adoption and implementation outcomes of the INFA program, and likelihood of these interventions being delivered long-term and scaled-up. Secondly, the investigators will evaluate the selected implementation strategies in action by examining adoption and fidelity, and also identify the CFIR determinants that influence these implementation outcomes. This will be done through FGDs/IDIs with the nursing leadership, programme implementers, and older adults. Additionally, the logic model and theory of change will be refined.

ELIGIBILITY:
Inclusion Criteria [Pre-implementation]:

1. Participants are healthcare professionals (nurses, doctors, allied health workers, nursing/clinical leadership) who are involved in the conceptualisation, implementation and/or delivery of the INFA programme.
2. They are able to share their views on the anticipated barriers and facilitators of implementing and delivering the INFA programme.
3. They consent to participating in the focus group discussion or in-depth interview.

Exclusion Criteria [Pre-implementation]:

* They do not consent to participating.

Inclusion Criteria [Implementation]:

1. Participants are 65 years or older
2. Has a Clinical Frailty Scale (CFS) rating of 4-6
3. Admitted to surgical and general medical wards

Exclusion Criteria [Implementation]:

1. All elective admissions
2. Individuals admitted from nursing or sheltered homes
3. Patients who are admitted for less than 48 hours.

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
[Implementation phase] Effectiveness of INFA Program - Functional status | Upon discharge and 6-months post-discharge
  It is hypothesized that with the implementation of the INFA program will lead to improved ADL functions.
  Changes in functional status will be measured using the modified Barthel Index of Activities of Daily Living (ADL) functional ability by comparing participants receiving INFA intervention on top of standard care, compared to participants who received only standard care.
[Implementation phase] Effectiveness of INFA Program - Implementation Strategies | Within 6 months post discharge
  To understand the effectiveness of the selected implementation strategies from the pre-implementation phase, qualitative interviews will be conducted on INFA implementors to understand the adoption, feasibility, sustainability, and scalability of the INFA program.

SECONDARY OUTCOMES:
[Implementation phase] Participant healthcare utilization | Upon discharge and 6-months post-discharge
  To compare the effectiveness of the INFA programme by analyzing data on participant's healthcare utilization such as number of unplanned hospital readmissions, Emergency Department visits and length-of-stay.
  Where possible, hospital data will be accessed to obtain the relevant data for analysis.
[Implementation phase] Health-Related Quality of Life (HRQoL) | Upon discharge and 6 months post-discharge.
  HRQoL will be measured using the five-level version of the EuroQoL 5 dimensions (EQ-5D-5L) instrument. Quality-Adjusted Life Years (QALYs) will be the primary measure of health benefits gained.
  Where possible, hospital data will be accessed to obtain the relevant data for analysis.
  Else, surveying of the participant's caregiver would be done.
[Implementation phase] Cost Effectiveness Analysis | 6 months prior to index admission and 6 months post-discharge
  The cost of providing the entire programme at a per patient level will be determined.
  This will include the cost of providing (1) INFA, (2) Nurse-led protocols, (3) GeriCARE and geriatricians referrals, (4) Discharge and follow-up planning.
  Where possible, hospital data will be accessed to obtain the relevant data for analysis.
  Else, surveying of the participant's caregiver would be done.

OTHER OUTCOMES:
[Implementation phase] INFA Process Indicators | Regular 1-month intervals after implementation phase have begun
  Guided by the developed logic model, relevant process indicators such as percentage of INFA assessments completed, proportion (%n) of eligible patients with nursing care plans initiated for applicable INFA domains, number of (actualized) referrals for each INFA domain, etc., will be collected to identify the implementation effectiveness of INFA program.
  Where possible, hospital data will be accessed to obtain the relevant data for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Chew, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singpaore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Background] Damschroder LJ, Reardon CM, Opra Widerquist MA, Lowery J. Conceptualizing outcomes for use with the Consolidated Framework for Implementation Research (CFIR): the CFIR Outcomes Addendum. Implement Sci. 2022 Jan 22;17(1):7. doi: 10.1186/s13012-021-01181-5. PMID 35065675
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Rezaei-Shahsavarloo Z, Atashzadeh-Shoorideh F, Gobbens RJJ, Ebadi A, Ghaedamini Harouni G. The impact of interventions on management of frailty in hospitalized frail older adults: a systematic review and meta-analysis. BMC Geriatr. 2020 Dec 3;20(1):526. doi: 10.1186/s12877-020-01935-8. PMID 33272208